CLINICAL TRIAL: NCT06101810
Title: Self-esteem in a General Psychiatric Population: Comparing Competitive Memory Training (COMET) and Cognitive Behavioral Therapy (CBT)
Brief Title: The Efficacy of Treatments to Improve Self-esteem
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: GGZ Noord-Holland-Noord (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GGZNHN23EJ
Record Dates: First submitted 2023-08-14; First posted 2023-10-26 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Self Esteem

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- COMET (Korrelboom) (Experimental): Korrelbooms' Competitive Memory Training (2011) (abbreviated COMET) is a cognitive behavioral therapy based on counter-conditioning. It uses positive self-verbalizations, imagination, posture and facial expression and music in a protocolized intervention consisting of 8 weekly group sessions of 90 minutes. For this study the protocol is extended with 1 session, to 9 sessions, in concertation with the author.
  Interventions: Behavioral: COMET
- CBT (De Neef) (Experimental): The cognitive behavioural protocol by De Neef (2010; 2018) has not been specifically named but is commonly referred to as 'the whitebook method' or 'cognitive behavioral therapy' (CBT). For convenience, this intervention will be addressed to as CBT in the current study.
  This intervention relies heavily on positive data logging to specifically focus on evidence that is contradictory to the negative core belief. Patients keep a positive data log (the 'whitebook') to write down positive events and positive qualities of themselves to achieve cognitive bias modification. They also receive psycho-education and practice on alternative behavior such as receiving compliments (which is also regarded as exposure), lowering perfectionist behavior and receiving criticism. In this protocolized intervention patients receive 9 to 11 weekly group sessions of 90 minutes. for this study a version of the protocol with 9 sessions is used.
  Interventions: Behavioral: CBT

INTERVENTIONS:
Behavioral: COMET — information already included in arm/group descriptions.
  Arms: COMET (Korrelboom)
Behavioral: CBT — information already included in arm/group descriptions.
  Arms: CBT (De Neef)

SUMMARY:
The goal of this study is to examine the effectivity of two self-esteem interventions (COMET (Korrelboom) and CBT (De Neef)) in a general psychiatric population.

The main questions it aims to answer are:

* is there a difference between the two interventions in effectiveness on increasing self-esteem?
* is there a difference between the two interventions in effect on levels of anxiety, depression and general mental health?
* are found effects on levels of anxiety, depression and general mental health associated with changes in self-esteem?
* is the ability to use imagination a moderator for outcomes in both conditions?

Participants are randomised over both conditions. At baseline (T0), end of treatment (T1) and follow-up at 6 months (T2) several outcome measures are conducted, such as RSES, DASS and MHC-SF.

DETAILED DESCRIPTION:
In this study, the investigators will examine the effectivity of self-esteem interventions.

To achieve this goal, the primary aim of this study is to examine if there is a difference in effectiveness between two interventions that have shown to be effective in ameliorating levels of low self-esteem in previous studies (ie. COMET (Korrelboom) and CBT (De Neef)).

Secondly, the investigators would like to find out if self-esteem interventions have an effect on levels of depression, anxiety and general mental health. This would give us a better understanding of the role of self-esteem as a trans-diagnostic factor.

The final aim of this study is to find out if some patients might profit more from one intervention over the other. One of the main differences between both interventions is that COMET heavily relies on imagination techniques and CBT does not. It could be possible that the extend to which patients are able to profit from an intervention which relies on imagination, depends on the ability or vividness in which they are able to use imagery. In this study the investigators will investigate if the ability to use mental imagery has an effect on treatment effects.

Design - In this study, research questions will be answered using a randomized clinical trial. After inclusion, patients are randomly assigned to one of the two conditions: 9 weeks of COMET + (ongoing) TAU versus 9 weeks of CBT + (ongoing) TAU. After baseline assessment participants will be randomized.

Population - All participants are adult (aged 18-65) outpatients of the regional community mental health teams of GGZ Noord-Holland Noord, a large secondary mental health care centre in the Netherlands with several locations. These teams treat patients with serious and complex psychiatric problems with any DSM-5 diagnosis (except those with a primary diagnosis of drug or alcohol related disorders and those with severe learning disabilities).

Including criterium is a self-perceived low self-esteem established by both patient and caregiver by means of (consent to) referral for self-esteem treatment.

ELIGIBILITY:
Inclusion Criteria:

- A self-perceived low self-esteem established by both patient and caregiver by means of (consent to) referral for self-esteem treatment.

Exclusion Criteria:

* severe suicidality for which hospitalization or other forms of crisis care is necessary,
* acute psychosis,
* current manic episode,
* current alcohol or drug abuse,
* insufficient knowledge of the Dutch language,
* illiteracy
* being unable to identify at least one positive aspect of oneself, which does not need to be felt as convincing for the participant. The latter is an excluding criterium formulated by the COMET protocol.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Rosenberg self-esteem scale (RSES) | Baseline (T0), end of treatment (T1)(one week after the last intervention session), follow-up (T2 at 6 months)
  Rosenberg self-esteem scale assesses global selfesteem on a 10-item questionnaire, items to be answered on a 4-point Likert scale ranging from 0 (strongly agree) to 3 (strongly disagree). Total scores range from 0 up to 30, with higher scores indicating a higher global self-esteem.

SECONDARY OUTCOMES:
Depression Anxiety Stress Scale (DASS) | Baseline (T0), end of treatment (T1)(one week after the last intervention session), follow-up (T2 at 6 months)
  Depression Anxiety Stress Scale is a 42-item questionnaire with items rated on a 4-point Likert scale, ranging from 0 (never) to 3 (definitely or most of the time). The DASS consists of three subscales of 14 items: Depression, Anxiety and Stress. Total scores on the subscales range from 0 up to 42, with higher scores indicating a higher levels of distress.
Mental Health Continuum - Short Form (MHC-SF) | Baseline (T0), end of treatment (T1)(one week after the last intervention session), follow-up (T2 at 6 months)
  Mental Health Continuum - Short Form is a 14 item questionnaire with items to be rated on a 6-point Likert scale, ranging from 0 (never) to 5 (every day). Higher scores mean a better outcome. Total score intends to measure positive mental health as a distinct indicator of mental well-being. Three subscales are Emotional well-being (presence of positive feelings), Psychological well-being (positive functioning in individual life) and Social well-being (positive functioning in community life).
  Higher scores indicate more well-being.
Plymouth Sensory Imagery Questionnaire (PsiQ-NL-35) | Baseline (T0)
  Plymouth Sensory Imagery Questionnaire is a 35 item questionnaire. It assesses mental imagery vividness on 5 items for 7 modalities (i.e., vision, sound, smell, taste, touch, bodily sensation and emotion). Each of the 7 modalities have a heading such as 'imagine the smell of…', followed by 5 items such as 'a rose' or 'burning wood'. Items are to be rated on a 11-point scale (0-10), ranging from 0 (no image at all) to 10 (as vivid as real life).

OTHER OUTCOMES:
Demographics | Baseline (T0)
  Demographics
DSM-5 classifications | Baseline (T0)
  Classifications according to the Diagnostic and Statistical Manual of Mental Disorders-5 (DSM-5)
Medication (type) | Measured from start of treatment until end of treatment (T1)(one week after the last intervention session), and from end of treatment (T1)(one week after the last intervention session) until follow-up (T2 at 6 months)
  Type of medication
Medication (dose) | Measured from start of treatment until end of treatment (T1)(one week after the last intervention session), and end of treatment (T1)(one week after the last intervention session) until follow-up (T2 at 6 months)
  Dose of medication per type of medication
Other forms of treatment | Measured from start of treatment until end of treatment (T1)(one week after the last intervention session), and from end of treatment (T1)(one week after the last intervention session) until follow-up (T2 at 6 months)
  Number of hours of other forms of treatment (Treatment As Usual/TAU) over the previous period.

CONTACTS AND LOCATIONS:
Overall Officials: Eva Velthorst, PhD, Principal Investigator — GGZ-NHN
Locations (1):
- Stichting GGZ Noord-Holland-Noord, Heerhugowaard, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No